CLINICAL TRIAL: NCT00000609
Title: Sudden Cardiac Death in Heart Failure Trial (SCD-HeFT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 112; U01HL055766 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2005-11

CONDITIONS: Arrhythmia; Cardiovascular Diseases; Death, Sudden, Cardiac; Heart Diseases; Heart Failure, Congestive; Heart Failure
MeSH Terms: conditions — Arrhythmias, Cardiac; Cardiovascular Diseases; Death, Sudden, Cardiac; Heart Diseases; Heart Failure | interventions — Amiodarone; Defibrillators, Implantable

INTERVENTIONS:
Drug: amiodarone
Device: defibrillators, implantable

SUMMARY:
To compare conventional treatment of congestive heart failure (CHF) with two experimental interventions: amiodarone and an implantable cardioverter-defibrillator (ICD).

DETAILED DESCRIPTION:
BACKGROUND:

Congestive heart failure is a major cause of mortality and morbidity, and sudden arrhythmic death is the cause of death in from 30 to 50 percent of those who die. The study addresses the problem and tests two interventions that have promise of benefit. To date, many of the therapies that have been tested for congestive heart failure have either been ineffective or actually decreased survival. Conventional therapy is still relatively ineffective in that recent studies such as the Congestive Heart Failure - Survival Trial of Antiarrhythmic Therapy (CHF-STAT) have demonstrated a mortality of 40 percent during two-and-half years of follow-up. The implantable cardioverter-defibrillator appears to be effective in patients who are resuscitated from cardiac arrest, but until recently, the devices required a thoracotomy and had to be reserved for patients with the highest risk for sudden death. The newer transvenous devices with pectoral patches can now be considered for broader applications. Although there have been mixed results with amiodarone in patients with congestive heart failure, there is a general consensus that it could be effective in the proper subset of patients with congestive heart failure. A comparison of the optimal device and drug is appropriate for such a high risk population.

DESIGN NARRATIVE:

Three-armed, randomized, multicenter trial conducted at over 125 North American, Australian and New Zealand sites. Patients were enrolled over 2.5 years after being randomly assigned to amiodarone, matched placebo or an implantable cardiac defibrillator (ICD). Median follow-up was 45.5 months. All three arms used conventional therapy for heart failure and coronary artery disease (ACE inhibitors, lipid lowering and beta-blockers). The central hypothesis was that amiodarone or the ICD would improve survival compared to placebo. The primary outcome was the prevention of all-cause mortality. Secondary outcome measures included cardiac mortality and arrhythmic mortality, morbidity, quality of life, and incremental cost-effectiveness of the interventions.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
Patients with New York Heart Association class II or class III heart failure and ejection fraction less than or equal to 35%.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-05; Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Lee — Duke University

REFERENCES:
- [Background] Bardy GH, Lee KL, Mark DB, Poole JE, Packer DL, Boineau R, Domanski M, Troutman C, Anderson J, Johnson G, McNulty SE, Clapp-Channing N, Davidson-Ray LD, Fraulo ES, Fishbein DP, Luceri RM, Ip JH; Sudden Cardiac Death in Heart Failure Trial (SCD-HeFT) Investigators. Amiodarone or an implantable cardioverter-defibrillator for congestive heart failure. N Engl J Med. 2005 Jan 20;352(3):225-37. doi: 10.1056/NEJMoa043399. PMID 15659722
- [Background] Kadish A. Prophylactic defibrillator implantation--toward an evidence-based approach. N Engl J Med. 2005 Jan 20;352(3):285-7. doi: 10.1056/NEJMe048351. No abstract available. PMID 15659729
- [Derived] Reeder HT, Shen C, Buxton AE, Haneuse SJ, Kramer DB. Joint Shock/Death Risk Prediction Model for Patients Considering Implantable Cardioverter-Defibrillators. Circ Cardiovasc Qual Outcomes. 2019 Aug;12(8):e005675. doi: 10.1161/CIRCOUTCOMES.119.005675. Epub 2019 Aug 15. PMID 31412732
- [Derived] Upshaw JN, Konstam MA, Klaveren Dv, Noubary F, Huggins GS, Kent DM. Multistate Model to Predict Heart Failure Hospitalizations and All-Cause Mortality in Outpatients With Heart Failure With Reduced Ejection Fraction: Model Derivation and External Validation. Circ Heart Fail. 2016 Aug;9(8):e003146. doi: 10.1161/CIRCHEARTFAILURE.116.003146. PMID 27514751
- [Derived] Fishbein DP, Hellkamp AS, Mark DB, Walsh MN, Poole JE, Anderson J, Johnson G, Lee KL, Bardy GH; SCD-HeFT Investigators. Use of the 6-min walk distance to identify variations in treatment benefits from implantable cardioverter-defibrillator and amiodarone: results from the SCD-HeFT (Sudden Cardiac Death in Heart Failure Trial). J Am Coll Cardiol. 2014 Jun 17;63(23):2560-2568. doi: 10.1016/j.jacc.2014.02.602. Epub 2014 Apr 9. PMID 24727258
- [Derived] Chen J, Johnson G, Hellkamp AS, Anderson J, Mark DB, Lee KL, Bardy GH, Poole JE. Rapid-rate nonsustained ventricular tachycardia found on implantable cardioverter-defibrillator interrogation: relationship to outcomes in the SCD-HeFT (Sudden Cardiac Death in Heart Failure Trial). J Am Coll Cardiol. 2013 May 28;61(21):2161-8. doi: 10.1016/j.jacc.2013.02.046. Epub 2013 Mar 26. PMID 23541974
- [Derived] Al-Khatib SM, Hellkamp A, Bardy GH, Hammill S, Hall WJ, Mark DB, Anstrom KJ, Curtis J, Al-Khalidi H, Curtis LH, Heidenreich P, Peterson ED, Sanders G, Clapp-Channing N, Lee KL, Moss AJ. Survival of patients receiving a primary prevention implantable cardioverter-defibrillator in clinical practice vs clinical trials. JAMA. 2013 Jan 2;309(1):55-62. doi: 10.1001/jama.2012.157182. PMID 23280225
- [Derived] Strauss DG, Poole JE, Wagner GS, Selvester RH, Miller JM, Anderson J, Johnson G, McNulty SE, Mark DB, Lee KL, Bardy GH, Wu KC. An ECG index of myocardial scar enhances prediction of defibrillator shocks: an analysis of the Sudden Cardiac Death in Heart Failure Trial. Heart Rhythm. 2011 Jan;8(1):38-45. doi: 10.1016/j.hrthm.2010.09.071. Epub 2010 Sep 25. PMID 20884379
- [Derived] Packer DL, Prutkin JM, Hellkamp AS, Mitchell LB, Bernstein RC, Wood F, Boehmer JP, Carlson MD, Frantz RP, McNulty SE, Rogers JG, Anderson J, Johnson GW, Walsh MN, Poole JE, Mark DB, Lee KL, Bardy GH. Impact of implantable cardioverter-defibrillator, amiodarone, and placebo on the mode of death in stable patients with heart failure: analysis from the sudden cardiac death in heart failure trial. Circulation. 2009 Dec 1;120(22):2170-6. doi: 10.1161/CIRCULATIONAHA.109.853689. Epub 2009 Nov 16. PMID 19917887
- [Derived] Levy WC, Lee KL, Hellkamp AS, Poole JE, Mozaffarian D, Linker DT, Maggioni AP, Anand I, Poole-Wilson PA, Fishbein DP, Johnson G, Anderson J, Mark DB, Bardy GH. Maximizing survival benefit with primary prevention implantable cardioverter-defibrillator therapy in a heart failure population. Circulation. 2009 Sep 8;120(10):835-42. doi: 10.1161/CIRCULATIONAHA.108.816884. Epub 2009 Aug 24. PMID 19704100
- [Derived] Olshansky B, Poole JE, Johnson G, Anderson J, Hellkamp AS, Packer D, Mark DB, Lee KL, Bardy GH; SCD-HeFT Investigators. Syncope predicts the outcome of cardiomyopathy patients: analysis of the SCD-HeFT study. J Am Coll Cardiol. 2008 Apr 1;51(13):1277-82. doi: 10.1016/j.jacc.2007.11.065. PMID 18371559